CLINICAL TRIAL: NCT01007435
Title: A Multi-center, Randomized, Double-blind, Parallel Group Study of the Safety, Disease Remission and Prevention of Structural Joint Damage During Treatment With Tocilizumab (TCZ), as a Monotherapy and in Combination With Methotrexate (MTX), Versus Methotrexate in Patients With Early, Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study of Tocilizumab as Monotherapy and in Combination With Methotrexate Versus Methotrexate in Patients With Early Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA19926; 2009-012759-12
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- (A) Tocilizumab 8 mg/kg + placebo to methotrexate (Experimental): Patients received tocilizumab 8 mg/kg iv every 4 weeks + placebo to methotrexate orally once a week for 104 weeks.
  Interventions: Drug: Tocilizumab; Drug: Placebo to methotrexate
- (B) Tocilizumab 8 mg/kg + methotrexate (Experimental): Patients received tocilizumab 8 mg/kg iv every 4 weeks + methotrexate orally once a week for 104 weeks.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate
- (C) Tocilizumab 4 mg/kg + methotrexate (Experimental): Patients received tocilizumab 4 mg/kg iv every 4 weeks + methotrexate orally once a week for 104 weeks.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate
- (D) Placebo to tocilizumab + methotrexate (Active Comparator): Patients received placebo tocilizumab intravenously (iv) every 4 weeks + methotrexate orally once a week for 104 weeks.
  Interventions: Drug: Placebo to tocilizumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab was supplied in vials.
  Other Names: RoActemra; Actemra
  Arms: (A) Tocilizumab 8 mg/kg + placebo to methotrexate; (B) Tocilizumab 8 mg/kg + methotrexate; (C) Tocilizumab 4 mg/kg + methotrexate
Drug: Placebo to tocilizumab — Placebo to tocilizumab was supplied in vials.
  Arms: (D) Placebo to tocilizumab + methotrexate
Drug: Methotrexate — Initially, patients received methotrexate 7.5 mg (3, 2.5 mg tablets) orally once a week. If a patient had swollen or tender joints, the dose was increased to 15 mg and 20 mg weekly, at the Week 4 and Week 8 visits, respectively.
  Arms: (B) Tocilizumab 8 mg/kg + methotrexate; (C) Tocilizumab 4 mg/kg + methotrexate; (D) Placebo to tocilizumab + methotrexate
Drug: Placebo to methotrexate — Patients received placebo to methotrexate orally once a week.
  Arms: (A) Tocilizumab 8 mg/kg + placebo to methotrexate

SUMMARY:
This randomized, double-blind, parallel group study will assess the safety, disease remission, and prevention of structural joint damage in patients with early moderate to severe rheumatoid arthritis treated with tocilizumab as monotherapy or in combination with methotrexate, versus methotrexate alone. Patients will be randomized to receive either (A) tocilizumab (8 mg/kg iv every 4 weeks) plus placebo, (B) tocilizumab (8 mg/kg iv every 4 weeks) plus methotrexate (7.5-20 mg po weekly), (C) tocilizumab (4 mg/kg iv every 4 weeks) plus methotrexate (7.5-20 mg po weekly), or (D) placebo plus methotrexate (7.5-20 mg po weekly). Patients in groups C and D who have not achieved low disease activity at week 52 can receive tocilizumab 8 mg/kg iv every 4 weeks. Anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Rheumatoid arthritis of ≤ 2 years duration.
* Disease Activity Score 28 (DAS28) > 3.2.
* Swollen joint count (SJC) ≥ 4 of 66 joints, tender joint count (TJC) ≥ 6 of 68 joints.
* Rheumatoid factor (RF) and/or anti-cyclic citrullinated peptide (anti-CCP) positive (if RF and anti-CCP negative > 1 erosion required at screening).
* Erythrocyte sedimentation rate (ESR) ≥ 28 mm/h or C-reactive protein (CRP) ≥ 10 mg/L at screening.

Exclusion Criteria:

* Previous treatment with tocilizumab.
* Previous treatment with methotrexate or biologic agent.
* Rheumatic autoimmune disease other than rheumatoid arthritis (RA).
* History of or current inflammatory joint disease other than RA.
* Functional class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2009-10-31 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2014-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (236):
- United States (61):
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Clnical & Translational Reseach Center for Alabama, PC, Tuscaloosa, Alabama
  - Arthrocare, Arthritis Care and Research, P.C., Mesa, Arizona
  - Sun Valley Arthritis Center, Peoria, Arizona
  - Talbert Medical Group, Huntington Beach, California
  - Uni of California - San Diego; Division of Rheumatology, La Jolla, California
  - Valerius Medical Group & Research Ctr of Greater Long Beach, Los Alamitos, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - San Diego Arthritis Med Clnc, San Diego, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Joao Nascimento, Bridgeport, Connecticut
  - New England Research Associates, Trumbull, Connecticut
  - Arthritis/Osteoporosis Treatment Center, Orange Park, Florida
  - Arthritis Center Palm Harbor, Palm Harbor, Florida
  - Arthritis Rsrch of Florida, Inc., Palm Harbor, Florida
  - Burnette & Silverfield, MDS, Tampa, Florida
  - Quad City Rheumatology, Sc, Moline, Illinois
  - Illinois Bone & Joint Inst., Morton Grove, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Physician'S Clinic of Iowa, Cedar Rapids, Iowa
  - Via Christi Clinic, PA, Wichita, Kansas
  - Baton Rouge Clinic, Amc, Baton Rouge, Louisiana
  - Osteoporosis & Clinical Trials Center, Cumberland, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Borgess Rheumatology, Kalamazoo, Michigan
  - Fiechtner Research Inc, Lansing, Michigan
  - Harbor Arthritis Center, Petoskey, Michigan
  - Park Nicollet Inst. ; Rtrc, Minneapolis, Minnesota
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - North Mississippi Medical Ctr; Internal Medicine Associates, Tupelo, Mississippi
  - Depaul Medical Group-SSM Healthcare, Florissant, Missouri
  - Dartmouth-Hitchcock Medical Center, Rheumatology 5C, Lebanon, New Hampshire
  - NJP Clinical Research, Clifton, New Jersey
  - Mark Fisher Md, Facr, Llc, Haddon Heights, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - Arthritis Health Associates; Clinical Research, Syracuse, New York
  - Asheville Arthritis & Osteoporosis Center, PA, Asheville, North Carolina
  - Durham Rheumatology, Durham, North Carolina
  - Ohio State University; Dept of Immunology, Columbus, Ohio
  - Southwest Rheumatology & Research Group, LLC, Middleburg Heights, Ohio
  - Health Research of Oklahoma, Llc, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - East Penn Rheumatology Associates, Pc, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Accurate Clinical Research, Houston, Texas
  - Houston Inst. For Clinical Research, Houston, Texas
  - Arthritis & Osteoporosis Associates, LLP, Lubbock, Texas
  - Texas Arthritis Research Center; Center for Arthritis & Rheumatic Diseases, San Antonio, Texas
  - Texas Research Center, Sugar Land, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
  - Arthritis Northwest, Spokane, Spokane, Washington
  - Tacoma Center For Arthritis Research, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
- Argentina (4):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Inst. de Rehabilitacion Psicofisica; Reumathology, Buenos Aires
  - Caici; Rheumatology, Rosario
  - Centro Medico Privado de Reumatologia; Reumathology, San Miguel
- Australia (6):
  - Royal Prince Alfred Hospital; Rheumatology, Camperdown, New South Wales
  - Sunshine Coast Rheumatology Research Unit, Maroochydore, Queensland
  - Queen Elizabeth Hospital; Rheumatology, Woodville, South Australia
  - Menzies Research Institute, Hobart, Tasmania
  - Cabrini Medical Centre; Rheumatology, Malvern, Victoria
  - Worthing Hospital, Murdoch, Western Australia
- Austria (3):
  - Lkh innsbruck - univ. Klinikum innsbruck - Tiroler landeskrankenanstalten ges.m.b.h.; Innere Medizin, Innsbruck
  - Kaiser Franz Josef Spital; Ii. Medizinische Abt., Vienna
  - Krankenhaus der stadt wien hietzing; ii. Med. Abt. / zentrum für rheumatologie, Vienna
- Brazil (8):
  - Centro Internacional de Pesquisa; Reumatologia, Goiânia, Goiás
  - Hospital das Clinicas - UFG;Reumatologia, Goiânia, Goiás
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras - CETI, Curtiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - PUCCamp; Reumatologia, Campinas, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP; Reumatologia, São Paulo, São Paulo
  - Centro Paulista de Investigacao Clinica - CEPIC, São Paulo, São Paulo
- Canada (14):
  - Arthritis Research Centre, Vancouver, British Columbia
  - Laurel Medical Clinic, Vancouver, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Nexus Clinical Research Centre, St. John's, Newfoundland and Labrador
  - Dr. William G. Bensen Medicine Professional Corporation, Hamilton, Ontario
  - K-W Musculoskeletal Research, Kitchener, Ontario
  - St. Joseph'S Health Care Centre; Rheumatology, London, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Niagara Peninsula Arthritis Centre, St. Catharines, Ontario
  - Hopital Maisonneuve- Rosemont; Rheumatology, Montreal, Quebec
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
  - Centre Re Recherche Saint-Louis, Québec
- China (4):
  - China-Japan Friendship Hospital, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
- Colombia (3):
  - Riesgo De Fractura; Rheumatology, Bogotá
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
  - Reumalab Sas; Rheumatology, Medellín
- Sjællands Universitetshospital, Køge; Reumatologisk Afdeling, Køge, Denmark
- Finland (2):
  - Helsinki University Central Hospital; Rheumatology Clinic, Helsinki
  - Kiljavan Lääketutkimus Oy, Hyvinkää
- France (7):
  - CH Jean Rougier; Rhumato Reed Fonctionnelle, Cahors
  - Fondation Hopital Saint Joseph; Rhumatologie, Marseille
  - Hopital Lapeyronie; Immunologie Rhumatologie, Montpellier
  - Hopital emile muller; Rhumatologie, Mulhouse
  - Hopital Porte Madeleine; Service de Rhumatologie, Orléans
  - Ch Pitie Salpetriere; Rhumatologie, Paris
  - Hopital Purpan; Rhumatologie, Toulouse
- Germany (15):
  - Kerckhoff-Klinik; Rheumatologie&klin.Immunologie, Bad Nauheim
  - Rheuma-Zentrum Baden-Baden Gmbh; Klinik Für Innere Medizin-Rheumatologie, Baden-Baden
  - Campus Charité Mitte Charité Centrum 12. Med.Klinik Abt.Rheumatologie u.Klin.Immunologie, Berlin
  - Schlosspark Klinik; Abt. Rheumatologie, Berlin
  - Klinik der Uni zu Köln; Klinik für Innere Medizin, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik III, Dresden
  - Dres. Florian Schuch, Ruediger de la Camp, Martin Hammerschmidt u.w., Erlangen
  - Schön Klinik Hamburg-Eilbek Klinik für Rheumatologie, Hamburg
  - Rheumapraxis PD Dr.med. Bernhard Heilig, Heidelberg
  - Rheumazentrum-Ruhrgebiet, St. Josefs-Krankenhaus; Rheumatologie, Herne
  - Gemeinschaftspraxis Dr. Von Hinueber/Dr. Demary; Rheumatologie, Hildesheim
  - Klinikum der Universität München; Bereich Pettenkoferstr.; Rheumaeinheit der medizinischen Klinik IV, München
  - Rheumapraxis an der Hase, Osnabrück
  - Evangelisches Fachkrankenhaus; Rheumaklinik, Ratingen
  - Universitätsklinikum Würzburg; Medizinische Klinik und Poliklinik II; Rheumatologie/Immunologie, Würzburg
- Greece (2):
  - Laiko General Hospital; Hematology Clinic, Athens
  - University General Hospital of Larissa; Rheumatology Unit, Larissa
- Guatemala (3):
  - Clinica Medica Del Dr Eduardo Alfredo Samayoa, Guatemala City
  - Private Practice, Guatemala City
  - Reuma-Centro, Guatemala City
- Hong Kong (3):
  - QUEEN MARY HOSPITAL; Division of Rheumatology & Clinical Immunology, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital; Department of Medicine, Hong Kong
  - Tuen Mun Hospital; Medicine & Geriatrics, Tuenmen
- Hungary (3):
  - Budai Irgalmasrendi Kórház KHT. II. Reumatológia, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum; Belgyógyászati Intézet, Reumatológiai Tanszék, Debrecen
  - Markhot Ferenc Hospital; Dep. of Rheumatology, Eger
- Ireland (3):
  - Cork Uni Hospital; Dept of Rheumatology, Cork
  - Adelaide and Meath Hospital; Rheumatology Department, Dublin
  - St.Vincent's University Hospital; Rheumatology Department, Dublin
- Israel (8):
  - Haemek Hospital; Rheumatology, Afula
  - Barzilai; Rheumatology, Ashkelon
  - Bnei Zion Medical Center; Rheumatology, Haifa
  - Hadassah University Hospital, Ein Karem; Rheumatology, Jerusalem
  - Hadassah Mount Scopus Hospital; Rheumatology, Jerusalem
  - Meir Medical Center; Internal Dept A, Kfar Saba
  - Chaim Sheba Medical Center; Rheumatology, Ramat Gan
  - Chaim Sheba Medical Center; Interna Dept B, Ramat Gan
- Italy (10):
  - Policlinico Universitario; Cattedra Di Reumatologia, Edificio 3, Napoli, Campania
  - Istituto Ortopedico Rizzoli; Unità di Reumatologia, Bologna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Reumatologia, Reggio Emilia, Emilia-Romagna
  - Campus Bio-Medico; Immunologia e Allergologia, Rome, Lazio
  - Policlinico Umberto I - Universita' La Sapienza ; Cattedra Di Reumatologia - Dept. Terapia Medica, Rome, Lazio
  - Università Degli Studi Di Genova - Dimi; Reumatologia, Genoa, Liguria
  - Ospedale Di Magenta Fornaroli; U.O. Di Reumatologia, Magenta, Lombardy
  - ASST FATEBENEFRATELLI SACCO; Reumatologia (Sacco), Milan, Lombardy
  - Ospedale S. Giovanni Bosco; S.C. A Direzione Uni Ria Di Immunologia Clinica, Turin, Piedmont
  - Policlinico Universitario Di Cagliari, Monserrato, Sardinia
- Mexico (8):
  - Centro de Investigación de Tratamientos Innovadores de Sinaloa (CITI), Culiacán, Sinaloa
  - Centro de Estudios de Investigacion Basica Y Clinica S.C.; Reumatologia, Guadalajara
  - Unidad de Reumatologia Rehabilitacion Integral; Centro Medico Del Angel, Mexicali
  - Unidad De Enfermedades; Cronico Degenerativas, SC., México
  - Cliditer SA de CV, Miexico City
  - Centro de Investigación Clínica de Morelia, S.C.; Reumatologia, Morelia
  - Hospital Universitario de Saltillo, Saltillo
  - Unidad de Enfermedades Reumaticas y Cronicodegenerativas, Torreón
- New Zealand (3):
  - North Shore Hospital, STAR Unit; Rheumatology Department, Auckland
  - Waikato Hospital; Rheumatology Outpatients, Hamilton
  - Timaru Hospital, Timaru
- Clinic of Rheumatology; Clinical Centre Skopje, Skopje, North Macedonia
- Centro de Infusion Marbella; Consultorios Royal Center Num 214, Panama City, Panama
- Peru (3):
  - Centro especializado de rehabilitacion fisica y del dolor cerfid - unidad de inv. En reumatologia, Lima
  - Abk Reuma Srl- Medicentro, Lima
  - Centro de Investigaciones Medicas/Hospital Maria Auxiliadora, San Juán de Miraflores
- Philippines (3):
  - Philippine General Hospital; Rheumatology, Manila
  - Jose Reyes Memorial Medical Center, Manila
  - Uni of Santo Tomas Hospital; Rheumatology, Manila
- Poland (6):
  - Szpital Specjalistyczny Nr 1; Oddzial Reumatologii I Rehabilitacji, Bytom
  - Wojewodzki Szpital Zespolony; Oddzial Reumatologii, Elblag
  - NZOZ REUMED Sp. z o.o., Lublin
  - Medyczne Centrum Hetmanska; Indywidualna Specjalistyczna Praktyka Lekarska, Poznan
  - Klinika Reumatologii I Chorób Wewn. Pum W Szczecinie; Samodzielny Publiczny Szpital Kliniczny Nr 1, Szczecin
  - Instytut Reumatologii im. Prof. Dr hab. Eleonory Reicher; Oddzial Wczesnej Diagnostyki Stawow, Warsaw
- Portugal (3):
  - HUC; Servico de Reumatologia, Coimbra
  - Hospital de Santa Maria; Servico de Reumatologia, Lisbon
  - Hospital de Sao Joao; Servico de Reumatologia, Porto
- Ponce School of Medicine; Caimed Center, Ponce, Puerto Rico
- Russia (12):
  - FSBI "National medico-surgical Centre n.a. N.I. Pirogov" of the Ministry of Healthcare, Moscow
  - FSBI "Scientific Research Institute of Rheumatology" of russian Academy of Medical Sciences, Moscow
  - FSBI "FSCC of particularized sorts of medical care and medical technologies of FMBA", Moscow
  - SBIH of Moscow "City clinical hospital #1 n.a. N.I. Pirogov" of Moscow Healthcare Department, Moscow
  - SBIH of Moscow "City Clinical Hospital #20 of Moscow Healthcare Department", Moscow
  - Ryazan State Medical University Named after I.P.Pavlov, Ryazan
  - SBEI of HPE "Northwestern State Medical University n.a. I.I.Mechnikov" of MoH of RF, Saint Petersburg
  - State institution of healthcare "Regional hospital for war veterans", Saratov
  - State Institution of Healthcare of Tula Region "Tula Regional Clinical Hospital", Tula
  - Budget Institution of Healthcare of Voronezh Region "Voronezh Regional Clinical Hospital #1", Voronezh
  - State Institution of Healthcare of Yaroslavl Region Clinical Hospital #8, Yaroslavl
  - Municipal Autonomous Institution of Healthcare "City Clinical Hospital #40", Yekaterinburg
- National University Hospital; Dept of Medicine, Singapore, Singapore
- South Africa (5):
  - Netcare Private Hospital, Bloemfontein
  - St Augustines Hospital; Rheumatology, Durban
  - Greenacres Hospital, Port Elizabeth
  - Clinical Research Unit, Pretoria
  - Winelands Research Centre, Stellenbosch
- Spain (10):
  - Hospital de Merida ;Servicio de Reumatologia, Mérida, Badajoz
  - Hospital Universitario Marques de Valdecilla; Servicio de Reumatologia, Santander, Cantabria
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Reumatologia, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Infanta Sofia; Servicio de Reumatologia, San Sebastián de los Reyes, Madrid
  - Hospital Univ. Central de Asturias; Servicio de Reumatologia, Oviedo, Principality of Asturias
  - Hospital Universitario Reina Sofia; Servicio de Reumatologia, Córdoba
  - Hospital General Universitario de Guadalajara; Servicio de Reumatologia, Guadalajara
  - Hospital Universitario de la Princesa; Servicio de Reumatologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Reumatologia, Seville
  - Hospital Univ. Nuestra Señora de Valme; Servicio de Reumatologia, Seville
- Sweden (2):
  - Karolinska University Hospital, Huddinge; Rheumatology, Huddinge
  - Karolinska Sjukhuset; Reumatologkliniken D2-1, Stockholm
- Thailand (4):
  - Chulalongkorn Hospital; Division of Rheumatology - Medicine, Bangkok
  - Phramongkutklao Hospital; Dept. of Medicine, Rheumatology, Bangkok
  - Ramathibodi Hospital, Mahidol Uni ; Allergy, Immunology & Rheumatology, Dept of Medicine, Bangkok
  - Songklanagarind Hospital; Department of Internal Medicine, Division of Rheumatology, Songkhla
- Iu Cerrahpasa Tip Fakultesi Ic Hastaliklari Anabilim Dali; Romatoloji Bilim Dali, Istanbul, Turkey (Türkiye)
- United Kingdom (12):
  - Addenbrooke'S Hospital; Rheumatology Research Unit, Cambridge
  - Cannock Chase Hospital; Rheumatology, Cannock
  - Royal Derby Hospital, Derby
  - Russells Hall Hospital; Rheumatology Department, Dudley
  - Maidstone Hospital; Dept of Rheumatology, Maidstone
  - Trafford General Hospital; Rheumatology, Manchester
  - Arrowe Park Hospital; Rheumatology Dept, Metropolitan Borough of Wirral
  - Royal Victoria Infirmary; Clinical Research Facility, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Royal Hallamshire Hospital; Rheumatology, Sheffield
  - Haywood Hospital; Staffordshire Rheumatology Centre, Stoke-on-Trent
  - Torbay Hospital; Dept of Rhematology, Torquay

REFERENCES:
- [Derived] Burmester GR, Rigby WF, van Vollenhoven RF, Kay J, Rubbert-Roth A, Blanco R, Kadva A, Dimonaco S. Tocilizumab combination therapy or monotherapy or methotrexate monotherapy in methotrexate-naive patients with early rheumatoid arthritis: 2-year clinical and radiographic results from the randomised, placebo-controlled FUNCTION trial. Ann Rheum Dis. 2017 Jul;76(7):1279-1284. doi: 10.1136/annrheumdis-2016-210561. Epub 2017 Apr 7. PMID 28389552
- [Derived] Burmester GR, Rigby WF, van Vollenhoven RF, Kay J, Rubbert-Roth A, Kelman A, Dimonaco S, Mitchell N. Tocilizumab in early progressive rheumatoid arthritis: FUNCTION, a randomised controlled trial. Ann Rheum Dis. 2016 Jun;75(6):1081-91. doi: 10.1136/annrheumdis-2015-207628. Epub 2015 Oct 28. PMID 26511996

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five of 1162 randomized patients (2 placebo to tocilizumab + methotrexate, 2 tocilizumab 4 mg/kg + methotrexate, 1 tocilizumab 8 mg/kg + methotrexate) did not receive any study treatment and were excluded from all analysis populations.
Groups:
- Placebo to Tocilizumab + Methotrexate: Patients received placebo tocilizumab intravenously (iv) every 4 weeks + methotrexate orally once a week for 104 weeks.
- Tocilizumab 4 mg/kg + Methotrexate: Patients received tocilizumab 4 mg/kg iv every 4 weeks + methotrexate orally once a week for 104 weeks.
- Tocilizumab 8 mg/kg + Methotrexate: Patients received tocilizumab 8 mg/kg iv every 4 weeks + methotrexate orally once a week for 104 weeks.
- Tocilizumab 8 mg/kg + Placebo to Methotrexate: Patients received tocilizumab 8 mg/kg iv every 4 weeks + placebo to methotrexate orally once a week for 104 weeks.
Period: Overall Study
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Started | 289 | 290 | 291 | 292
Completed | 226 | 231 | 227 | 236
Not Completed | 63 | 59 | 64 | 56
Not completed — Adverse Event | 16 | 25 | 47 | 31
Not completed — Death | 2 | 4 | 2 | 1
Not completed — Insufficient Therapeutic Response | 21 | 7 | 2 | 9
Not completed — Violation of Selection Criteria at Entry | 3 | 5 | 2 | 0
Not completed — Other Protocol Violation | 2 | 0 | 1 | 0
Not completed — Refused Treatment | 13 | 13 | 5 | 8
Not completed — Failure to Return | 5 | 4 | 3 | 6
Not completed — Reason not Specified | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were based on the intent-to-treat (ITT) population. Five of 1162 randomized patients (2 placebo + methotrexate, 2 tocilizumab 4 mg/kg + methotrexate, 1 tocilizumab 8 mg/kg + methotrexate) did not receive any study treatment and were excluded from all analysis populations. The ITT population therefore included 1157 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate | Total
Number analyzed (Participants) | 287 | 288 | 290 | 292 | 1157
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (13.10) | 51.2 (13.84) | 49.5 (13.70) | 49.9 (13.22) | 50.1 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 228 | 228 | 219 | 904
  Male | 58 | 60 | 62 | 73 | 253

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Disease Activity Score 28 (DAS28) Remission Response at Week 24
Description: A participant has a DAS28 remission response if their DAS28 < 2.6. The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Week 24
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 287 | 288 | 290 | 292
Percentage of participants | 15.0 [10.9 to 19.1] | 31.9 [26.6 to 37.3] | 44.8 [39.1 to 50.6] | 38.7 [33.1 to 44.3]
Statistical Analysis 1: Comparison: Placebo to Tocilizumab + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; The null hypothesis is that there is no difference in the DAS28 remission response at Week 24 between the placebo to tocilizumab + methotrexate and the tocilizumab 8 mg/kg + methotrexate treatment groups; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A hierarchy of statistical testing was implemented in order to control the type I error rate for multiple comparisons; The stratification factors, region and serologic status, were included in the model; Odds Ratio (OR) = 4.77, 95% CI 2-sided [3.19 to 7.14] — Last observation carried forward was used for TJC and SJC. No imputation was used for ESR and GH. Patients who withdrew prematurely or where a DAS28 could not be calculated were set to "non-responder"
Statistical Analysis 2: Comparison: Placebo to Tocilizumab + Methotrexate vs Tocilizumab 8 mg/kg + Placebo to Methotrexate; The null hypothesis is that there is no difference in the DAS28 remission response at Week 24 between the placebo to tocilizumab + methotrexate and the tocilizumab 8 mg/kg + placebo to methotrexate treatment groups; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A hierarchy of statistical testing was implemented in order to control the type I error rate for multiple comparisons; The stratification factors, region and serologic status, were included in the model; Odds Ratio (OR) = 3.70, 95% CI 2-sided [2.47 to 5.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo to Tocilizumab + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; The null hypothesis is that there is no difference in the DAS28 remission response at Week 24 between the placebo to tocilizumab + methotrexate and the tocilizumab 4 mg/kg + methotrexate treatment groups; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A hierarchy of statistical testing was implemented in order to control the type I error rate for multiple comparisons. This comparison came after the break in statistical hierarchy; The stratification factors, region and serologic status, were included in the model; Odds Ratio (OR) = 2.72, 95% CI 2-sided [1.80 to 4.11] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With a Disease Activity Score 28 (DAS28) Remission Response at Week 52
Time Frame: Week 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 287 | 288 | 290 | 292
Percentage of participants | 19.5 | 34.0 | 49.0 | 39.4

3. Secondary Outcome: Percentage of Patients With an Improvement ≥ 20%, 50%, or 70% in American College of Rheumatology (ACR) Score (ACR20/50/70) From Baseline to Weeks 24 and 52
Description: Improvement must be seen in tender (68) and swollen (66) joint counts. Joints were assessed and classified as swollen/not swollen and tender/not tender by pressure and joint manipulation. Improvement must also be seen in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, the extreme left end of the line "no disease activity" [symptom-free and no arthritis symptoms] and the extreme right end "maximum disease activity"; patient assessment of pain in previous the 24 hours on a VAS (extreme left end of the line "no pain" and the extreme right end "unbearable pain"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C-reactive protein (CRP), or erythrocyte sedimentation rate if CRP was missing.
Time Frame: Baseline to Weeks 24 and 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 287 | 288 | 290 | 292
Percentage of participants
  Week 24: ACR 20 | 65.2 | 73.6 | 74.5 | 70.2
  Week 24: ACR 50 | 43.2 | 47.9 | 56.9 | 47.6
  Week 24: ACR 70 | 25.4 | 34.7 | 38.6 | 30.1
  Week 52: ACR 20 | 57.1 | 62.8 | 67.2 | 63.0
  Week 52: ACR 50 | 40.8 | 52.4 | 55.9 | 49.3
  Week 52: ACR 70 | 28.9 | 37.2 | 43.1 | 36.0

4. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 52
Description: The mTSS is a measure of joint damage and includes measures of joint erosion (JE) and joint space narrowing (JSN). The JE score, using the van der Heijde modification, measures erosion severity in 32 hand joints and 12 foot joints. Each hand joint is scored from 0 to 5 and each foot joint is scored from 0 to 10; the total score ranges from 0 to 280. Each joint is scored according to the surface area involved. A score of 10 indicates extensive loss of bone from more than one-half of the articulating bone; a score of 0 indicates no erosion. The JSN score measures the severity of JSN in 30 hand joints (15 per hand) and 12 foot joints (6 per foot). Each joint, including subluxation, is scored from 0 to 4; the total score ranges from 0 to 168. A higher score indicates more joint space narrowing. The mTSS ranges from 0 to 448 (280+168). A higher mTSS score indicates greater damage. A negative change score indicates improvement.
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 267 | 267 | 273 | 275
Units on a scale | 1.14 (4.297) | 0.42 (2.929) | 0.08 (2.090) | 0.26 (1.876)

5. Secondary Outcome: Change From Baseline in Modified Sharp Erosion Score at Week 52
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 267 | 267 | 273 | 275
Units on a scale | 0.63 (2.556) | 0.25 (1.686) | 0.05 (1.736) | 0.15 (1.544)

6. Secondary Outcome: Change From Baseline in Sharp Joint Space Narrowing Score at Week 52
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 267 | 268 | 273 | 275
Units on a scale | 0.51 (2.362) | 0.17 (1.645) | 0.03 (0.751) | 0.11 (1.046)

7. Secondary Outcome: Percentage of Participants With a Major Clinical Response at Week 52
Description: A major clinical response is defined as an ACR70 response that is maintained for 6 consecutive months (24 weeks) for any 24-week period between Week 2 and Week 52.
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 287 | 288 | 290 | 292
Percentage of participants | 16 | 22 | 31 | 22

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Weeks 24 and 52
Description: The Stanford HAQ-DI is a patient completed questionnaire specific for rheumatoid arthritis. The HAQ-DI assesses how well the patient is able to perform 8 activities: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. The patient answers 20 questions with 1 of 4 responses with the past week as the time frame: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The highest score for any question in a category determines the category score. The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement.
Time Frame: Baseline to Weeks 24 and 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 287 | 288 | 290 | 292
Units on a scale
  Week 24 (n=246, 255, 250, 265) | -0.71 (0.718) | -0.92 (0.736) | -0.91 (0.695) | -0.82 (0.739)
  Week 52 (n=214, 227, 228, 230) | -0.76 (0.800) | -1.00 (0.795) | -0.97 (0.700) | -0.87 (0.776)

9. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Physical Component Summary (PCS) Scores at Weeks 24 and 52
Description: The SF-36 Health Survey (Version 2) is a standardized questionnaire consisting of 36 questions that measures patient-reported symptoms on 8 dimensions; it is used to assess health-related quality of life (HRQoL). The Physical Component Summary (PCS) score summarizes the subscales Physical Functioning, Role-Physical, Bodily Pain, and General Health. The Mental Component Summary (MCS) score summarizes the subscales Vitality, Social Functioning, Role-Emotional, and Mental Health. Each score was scaled from 0 to 100. A positive change score indicates better HRQoL.
Time Frame: Baseline to Weeks 24 and 52
Population: Intent-to-treat population: All randomized participants who received at least 1 tocilizumab/placebo infusion.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Number analyzed (Participants) | 287 | 288 | 290 | 292
Units on a scale
  Week 24 (n=237, 247, 246, 255) | 9.35 (9.763) | 11.33 (9.282) | 12.13 (9.263) | 10.75 (10.055)
  Week 52 (n=204, 225, 221, 224) | 10.72 (10.389) | 12.27 (10.509) | 13.52 (9.848) | 11.73 (10.691)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from Baseline through Week 52.
Description: Safety population: All patients who received at least 1 tocilizumab/placebo infusion and had at least 1 post-dose safety assessment. 7 patients were excluded from the safety population (no treatment received or no post-baseline safety data). The total safety population included 1153 patients.
Arm/Group | Placebo to Tocilizumab + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Placebo to Methotrexate
Serious Adverse Events (participants affected / at risk) | 24/282 | 29/289 | 31/290 | 25/292
Other Adverse Events (participants affected / at risk) | 177/282 | 182/289 | 201/290 | 163/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Tocilizumab + Methotrexate (N=282) | Tocilizumab 4 mg/kg + Methotrexate (N=289) | Tocilizumab 8 mg/kg + Methotrexate (N=290) | Tocilizumab 8 mg/kg + Placebo to Methotrexate (N=292)
Pneumonia (Infections and infestations) | 1 | 4 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 3 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 1
Pneumococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Oteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Tocilizumab + Methotrexate (N=282) | Tocilizumab 4 mg/kg + Methotrexate (N=289) | Tocilizumab 8 mg/kg + Methotrexate (N=290) | Tocilizumab 8 mg/kg + Placebo to Methotrexate (N=292)
Upper respiratory tract infection (Infections and infestations) | 40 | 37 | 30 | 39
Nasopharyngitis (Infections and infestations) | 38 | 40 | 28 | 27
Urinary tract infection (Infections and infestations) | 13 | 18 | 14 | 10
Bronchitis (Infections and infestations) | 6 | 18 | 20 | 8
Alanine aminotransferase increased (Investigations) | 29 | 39 | 55 | 22
Transaminases increased (Investigations) | 23 | 35 | 40 | 22
Aspartate aminotransferase increased (Investigations) | 8 | 8 | 17 | 11
Nausea (Gastrointestinal disorders) | 46 | 41 | 43 | 19
Diarrhoea (Gastrointestinal disorders) | 18 | 16 | 19 | 18
Dyspepsia (Gastrointestinal disorders) | 16 | 17 | 11 | 14
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 21 | 9 | 16 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 10 | 8 | 19
Hypertension (Vascular disorders) | 21 | 16 | 23 | 25
Headache (Nervous system disorders) | 12 | 20 | 18 | 20
Rash (Skin and subcutaneous tissue disorders) | 3 | 18 | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.